CLINICAL TRIAL: NCT00462228
Title: Double-blind Cross-over Study of the Effect of Namenda on Short Term Memory and Attention in Patients With Mild to Moderate Traumatic Brain Injury, Protocol NAM-MD-44
Brief Title: Effect of Namenda on Short Term Memory and Attention in Patients With Mild to Moderate Traumatic Brain Injury
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped due to a lack of additional subjects.
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NAM-MD-44
Record Dates: First submitted 2007-04-10; First posted 2007-04-18 (Estimated); Results first posted 2013-11-18 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2016-10

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; memory; attention
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memantine (Experimental): Subjects will be titrated up to 20 mg of memantine per day for 12 weeks, followed by placebo for 12 weeks
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): Subjects will be titrated up to 20 mg of placebo per day for 12 weeks, followed by memantine for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — After randomization of the subject, subjects will be titrated up to 20 mg of memantine or placebo per day. Memantine and placebo are provided as 5 mg tablets. Subjects will be started at 5 mg per day. The dose will be increased by 5 mg increments to 10 mg per day (5 mg twice per day), 15 mg per day (5 mg and 10 mg as separate doses) and 20 mg per day (10 mg twice per day). The minimum interval between dose increases will be one week. Subjects will take memantine or placebo for 12 weeks during each part of the crossover study. Subjects are randomized to begin either memantine or placebo in each arm of the study.
  Other Names: Namenda
  Arms: Memantine
Drug: Placebo — After randomization of the subject, subjects will be titrated up to 20 mg of memantine or placebo per day. Memantine and placebo are provided as 5 mg tablets. Subjects will be started at 5 mg per day. The dose will be increased by 5 mg increments to 10 mg per day (5 mg twice per day), 15 mg per day (5 mg and 10 mg as separate doses) and 20 mg per day (10 mg twice per day). The minimum interval between dose increases will be one week. Subjects will take memantine or placebo for 12 weeks during each part of the crossover study. Subjects are randomized to begin either memantine or placebo in each arm of the study.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether memantine (Namenda) improves memory and attention in patients with mild to moderate traumatic brain injury.

DETAILED DESCRIPTION:
Background and significance:

Each year in the United States approximately 1.5 million people sustain a traumatic brain injury (TBI) and of these approximately 80-90,000 result in long-term or lifelong disability. An estimated 5.3 million people are currently living with a disability due to TBI. The Centers for Disease Control (CDC) estimated that about 75% (1.1 million) of the reported TBIs are concussions or other forms of mild TBIs (MTBI). However, the incidence of MTBI has been vastly underestimated according to a CDC Report to Congress.

The long term problem associated with MTBI is primarily memory impairment. Memory impairment resulting form MTBI is not likely to improve with time beyond the initial stabilizing period of about one year post-injury. Dementia from Alzheimer's Disease produces cognitive problems that are similar to those experienced by patients with mild to moderate traumatic brain injury. The efficacy of Namenda for treatment of cognitive problems due to Alzheimer's Dementia suggests it may have efficacy for treatment of short term memory and attention deficits in patients with mild to moderate traumatic brain injury.

Overall Design and Plan of Study:

Twenty post-TBI patients whose TBI occurred at least 1 year prior to beginning the study will be recruited for this pilot study. Patients who meet screening criteria will have cognitive abilities assessed at baseline and at subsequent visits while taking Namenda or placebo. Patients will be randomly assigned to begin either Namenda or placebo and will then crossover to the alternate treatment. Each patient will participate in the study for a total of 32 to 34 weeks. Patients completing the study will have 10 total visits and 6 visits at which a cognitive test battery will be administered. This will include 24 weeks of study drug treatment (12 weeks of Namenda and 12 weeks of placebo) and two 4-week washout periods. Patients will be titrated up to 20 mg of Namenda per day. Namenda and placebo will be provided by Forest Laboratories Inc.

Cognitive screening criteria include a Galveston Orientation and Amnesia Test (GOAT) score of at least 75, and either a Mini-Mental State Exam (MMSE) score of 20 to 27 obtained at the screening visit, or a California Verbal Learning Test (CVLT) total score for trials 1-5 one standard deviation lower than the age matched normative score. The CVLT score for inclusion may be obtained from the medical record provided that the CVLT testing occurred one year or more post TBI and within two years of study entry.

The cognitive test battery measurements will be made at the first baseline before Namenda or placebo administration (week 0), and at weeks 6, & 12 after Namenda or placebo administration. After washout for 4 weeks, the second baseline (week 16) will be assessed, and the cognitive test battery will be administered again at weeks 22 & 28 after Namenda or placebo administration.

The cognitive test battery used to assess efficacy will utilize the following tests;

Verbal Memory: Hopkins Verbal Learning Test Revised (HVLT-R). Visual Memory: Brief VisuoSpatial Memory Test Revised (BVMT-R). Speed of processing: Trail Making Test Part A. Attention: Trail Making Test Part B. Memory/processing speed: Symbol Digit Modality Test (SDMT).

The primary endpoints for cognitive assessment will be the HVLT-R and the BVMT-R. The 6 different forms of the HVLT-R and BVMT-R will be administered at each of the 6 cognitive test battery assessments. The sequence of forms administered will be randomized. The other listed cognitive tests will be considered secondary endpoints. An additional secondary efficacy endpoint will be the Physicians Global Impression of Change which will be recorded with the same visit frequency as other cognitive tests.

In addition to the neuropsychological tests, patients will have physical examinations, electrocardiograms, and laboratory tests of blood and urine. Safety and tolerability will be monitored by clinical assessment, reporting of adverse events, and laboratory values. Patient health will be assessed at clinic visits every 3-6 weeks throughout the study. Serum pregnancy (for females of child bearing potential) will be completed at screening and at weeks 12 and 28. Urine pregnancy tests will be completed at baseline (week 0) and weeks 16 & 32. A Safety Officer will be utilized as the primary means of monitoring safety of the study. The Safety Officer will be a physician not associated with the study in any other capacity. The Safety Officer will be given periodic reports of clinical assessments, laboratory values, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will have persistent memory and attention deficits due to a closed traumatic brain injury not less than one year prior to entrance in the study.
2. Meet or exceed American Congress of Rehabilitation Medicine (ACRM) criteria for mild TBI.
3. Mini-Mental State Exam (MMSE) score of 20 to 27 at the screening visit or a California Verbal Learning Test (CVLT) score for trials 1-5 one standard deviation lower than the age matched normative score. The CVLT score from the medical record may be used for entry criteria if it was obtained one year or more post-TBI and within two years of study entry.
4. Galveston Orientation and Amnesia Test (GOAT) score of at least 75.
5. Be of sufficient cognitive ability to complete neuropsychological tests.
6. Male or female, 18-50 years of age.
7. Females of childbearing potential must use acceptable means of birth control and have a negative screening beta-human chorionic gonadotrophin (b-HCG) pregnancy test. Acceptable birth control includes hormonal birth control (such as oral birth control pills, implanted or injected contraceptives), an intrauterine device (IUD), surgical sterilization (such as tubal ligation or hysterectomy), a spermicide with barrier methods (condoms or diaphragm), or a partner who has had a vasectomy.
8. Patients taking donepezil (Aricept) or rivastigmine (Exelon) must be at a steady state dose for a minimum of six months.
9. Patients taking any other medication(s) affecting cognition must be at a steady state dose for a minimum of two months.
10. Able to provide written informed consent.
11. Able to read, write, and speak in English.
12. Willing and able to comply with the physician's instructions for all aspects of the study.

Exclusion Criteria:

1. Patients must not have any medical or psychiatric disorder that in the opinion of the PI would interfere with or bias the assessment of efficacy or place their health at risk when placed on the memantine (Namenda) regimen.
2. Patients with a history of seizure are excluded.
3. Patients with a history of severe renal insufficiency are excluded.
4. Patients must not have taken any experimental drug within the last 30 days prior to entering the protocol.
5. Patients must not have taken any drug known to have major organ system toxicity within the last 30 days prior to entering the protocol.
6. Women who are pregnant, nursing, or intend to become pregnant during the study are excluded.
7. Patients with a penetrating TBI are excluded.
8. Patients whose screening laboratory values are 1.5 times greater than upper limits of normal range(ULN) are excluded.
9. Patients with systolic blood pressure greater than 180 mm Hg or less than 90 mm Hg or diastolic blood pressure greater than 105 mm Hg or less than 50 mm Hg at the screening visit are excluded.
10. Concomitant use of amantadine (Symmetrel) is prohibited and a washout period of 4 weeks is required before study entry.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2007-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S. Jon Rupright, D.O., Principal Investigator — Associate Professer, Clinical Physical Medicine & Rehabilitation, School of Medicine, University of Missouri-Columbia; George R. Johnstone, Ph.D., Principal Investigator — Professor, Department of Health Psychology, University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by contacting patients of the principal investigator (PI) when they presented for regularly scheduled clinic appointments or by referrals from colleagues. The recruitment period was from was from July 2007 through December 2010.
Groups:
- Overall Study: All 11 baseline subjects completed the three periods of the study: memantine treatment, placebo treatment, and no treatment (washout period) in this crossover design. Five subjects were randomized to begin the study by taking memantine and crossover to placebo; seven subjects began with placebo and crossed over to memantine.
Period: Memantine or Placebo 12 Weeks
Arm/Group | Overall Study
Started | 11
Completed | 11
Not Completed | 0
Period: No Treatment (Washout) 4 Weeks
Arm/Group | Overall Study
Started | 11
Completed | 11
Not Completed | 0
Period: Placebo or Memantine 12 Weeks
Arm/Group | Overall Study
Started | 11
Completed | 11
Not Completed | 0
Period: No Treatment (Washout) 4 Weeks
Arm/Group | Overall Study
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All 11 baseline subjects completed the three periods of the study: memantine treatment, placebo treatment, and no treatment (washout period) in this crossover design.
Arm/Group | Overall Study
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (8.1)
Gender [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Improvements From Baseline Scores After 6 and 12 Weeks of Memantine Compared to Placebo on the Hopkins Verbal Learning Test Revised (HVLT-R) Total Recall Learning Scores.
Description: HVLT-R Learning Scores provide a brief assessment of immediate recall, delayed recall and delayed recognition. It is administered by reading the words aloud, then asking the client to verbally repeat the list of words (immediately; then after a delay), and identify the words from a word list that is presented verbally.
  The HVLT-R is easy to administer and score, and is well-tolerated by even significantly-impaired individuals. Tasks include three learning trials, which, when combined produce a total recall score; a delayed recall (25-30 minute delay) trial, and a yes/no delayed recognition trial. Raw scores are derived for Total Recall, Delayed Recall, Retention (percent retained) and a Recognition Discrimination Index.
  These results are for the HVLT-R total recall raw learning score. The HVLT-R total recall raw learning score ranges from 0 to 36 with 36 being the highest and best possible score.
Time Frame: Baseline, 6 weeks, and 12 weeks after beginning memantine or placebo
Population: All subjects completing the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Memantine: All subject scores for memantine regardless of sequence in the crossover design.
- Placebo: All subject scores for placebo regardless of sequence in the crossover design.
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 11 | 11
units on a scale
  baseline score | 20.91 (6.2) | 19.09 (3.7)
  6 week score | 19.09 (3.7) | 19.45 (4.2)
  12 week score | 19.73 (5.8) | 19.00 (4.2)
Statistical Analysis 1: Comparison: Memantine vs Placebo; Null hypothesis: The change from baseline occurring with memantine is equal to the change from baseline occurring with placebo at 6 weeks for HVLT-R total recall learning scores; Test type: Superiority or Other; p = 0.55, Sign test — 6 week comparison, alpha = 0.05
Statistical Analysis 2: Comparison: Memantine vs Placebo; Null hypothesis:The change from baseline occurring with memantine is equal to the change from baseline occurring with placebo at 12 weeks for HVLT-R total recall learning scores; Test type: Superiority or Other; p = 1.00, Sign test — 12 week comparison, alpha = 0.05
Statistical Analysis 3: Comparison: Memantine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.45, Wilcoxon (Mann-Whitney) — 6 week comparison, alpha = 0.05
Statistical Analysis 4: Comparison: Memantine vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.43, Wilcoxon (Mann-Whitney) — 12 week comparison, alpha = 0.05

2. Primary Outcome: Improvements From Baseline Scores After 6 and 12 Weeks of Memantine Compared to Placebo on the Hopkins Verbal Learning Test Revised (HVLT-R) Delayed Recall Scores.
Description: HVLT-R Learning Scores provide a brief assessment of immediate recall, delayed recall and delayed recognition. It is administered by reading the words aloud, then asking the client to verbally repeat the list of words (immediately; then after a delay), and identify the words from a word list that is presented verbally.
  The HVLT-R is easy to administer and score, and is well-tolerated by even significantly-impaired individuals. Tasks include three learning trials, which, when combined produce a total recall raw score; a delayed recall (25-30 minute delay) trial, and a yes/no delayed recognition trial. Raw scores are derived for Total Recall, Delayed Recall, Retention (percent retained) and a Recognition Discrimination Index.
  These scores are for the delayed recall learning raw score. The HVLT-R delayed recall raw score ranges from 0 to 12 with 12 being the highest and best possible score.
Time Frame: Baseline, 6 weeks, and 12 weeks after beginning memantine or placebo
Population: All subjects completing the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 11 | 11
units on a scale
  baseline score | 5.64 (3.8) | 4.36 (2.5)
  6 week score | 4.45 (2.7) | 5.18 (3.5)
  12 week score | 4.73 (3.3) | 5.82 (3.5)
Statistical Analysis 1: Comparison: Memantine vs Placebo; Null hypothesis: The change from baseline occurring with memantine is equal to the change from baseline occurring with placebo at 6 weeks for HVLT-R delayed recall scores; Test type: Superiority or Other; p = 0.23, Sign test — 6 week comparison,alpha = 0.05
Statistical Analysis 2: Comparison: Memantine vs Placebo; Null hypothesis: The change from baseline occurring with memantine is equal to the change from baseline occurring with placebo at 12 weeks for HVLT-R delayed recall scores; Test type: Superiority or Other; p = 0.022, Sign test — 12 week comparison, alpha = 0.05
Statistical Analysis 3: Comparison: Memantine vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.06, Wilcoxon (Mann-Whitney) — 6 week comparison, alpha = 0.05
Statistical Analysis 4: Comparison: Memantine vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.027, Wilcoxon (Mann-Whitney) — 12 week comparison, alpha = 0.05

3. Secondary Outcome: Improvements From Baseline Scores After 6 and 12 Weeks of Memantine Compared to Placebo on the Trail Making Test Part A.
Description: Trail Making Test Part A consists of 25 circles on a piece of paper with the numbers 1-25 written randomly in the circles. The test taker's task is to start with number one and draw a line from that circle to the circle with the number two in it to the circle with the three in it, etc. The person continues to connect the circles in numerical order until they reach number 25. Lower scores are better scores and the range of scores can be from 0 to no limit for Trail Making Test part A. This is a timed test and the number of seconds to complete the task is recorded.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 11 | 11
seconds
  baseline score | 49.5 (21.7) | 43.5 (13.8)
  6 week score | 48.1 (21.4) | 41.5 (13.6)
  12 week score | 40.5 (14.9) | 38.5 (12.6)
Statistical Analysis 1: Comparison: Memantine vs Placebo; Null hypothesis: The change from baseline occurring with memantine is equal to the change from baseline occurring with placebo at 6 weeks for the Trail Making Test Part A; Test type: Superiority or Other; p = 1.0, Sign test — 6 week comparison, alpha = 0.05
Statistical Analysis 2: Comparison: Memantine vs Placebo; Null hypothesis: The change from baseline occurring with memantine is equal to the change from baseline occurring with placebo at 12 weeks for the Trail Making Test Part A; Test type: Superiority or Other; p = 0.55, Sign test — 12 week comparison, alpha = 0.05
Statistical Analysis 3: Comparison: Memantine vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.81, Wilcoxon (Mann-Whitney) — 6 week comparison, alpha = 0.05
Statistical Analysis 4: Comparison: Memantine vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.57, Wilcoxon (Mann-Whitney) — 12 week comparison, alpha = 0.05

4. Secondary Outcome: Improvements From Baseline Scores After 6 and 12 Weeks of Memantine Compared to Placebo on the Trail Making Test Part B.
Description: Trail Making Test Part B consists of 24 circles on a piece of paper, but rather than all of the circles containing numbers, half of the circles have the numbers 1-12 in them and the other half (12) contain the letters A-L. The person taking the test has the more difficult task of drawing a line from one circle to the next in ascending order; however, he must alternate the circles with numbers in them (1-13) with circles with letters in them (A-L). In other words, he is to connect the circles in order like this: 1-A-2-B-3-C-4-D-5-E and so on. Lower scores are better scores and the range of scores can be from 0 to no limit for Trail Making Test part B. This is a timed test and the number of seconds to complete the task is recorded.
Time Frame: Baseline, 6 weeks, and 12 weeks after beginning memantine or placebo
Population: All subjects completing the study.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 11 | 11
seconds
  baseline score | 104.6 (54) | 113.3 (63)
  6 week score | 128.7 (94) | 100.8 (38)
  12 week score | 86.6 (32) | 105.5 (69)
Statistical Analysis 1: Comparison: Memantine vs Placebo; Null hypothesis: The change from baseline occurring with memantine is equal to the change from baseline occurring with placebo at 6 weeks for the Trail Making Test Part B; Test type: Superiority or Other; p = 0.55, Sign test — 6 week comparison, alpha = 0.05
Statistical Analysis 2: Comparison: Memantine vs Placebo; Null hypothesis: The change from baseline occurring with memantine is equal to the change from baseline occurring with placebo at 12 weeks for the Trail Making Test Part B; Test type: Superiority or Other; p = 1.0, Sign test — 12 week comparison, alpha = 0.05
Statistical Analysis 3: Comparison: Memantine vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.17, Wilcoxon (Mann-Whitney) — 6 week comparison, alpha = 0.05
Statistical Analysis 4: Comparison: Memantine vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.64, Wilcoxon (Mann-Whitney) — 12 week comparison, alpha = 0.05

5. Primary Outcome: Improvements From Baseline Scores After 6 and 12 Weeks of Memantine Compared to Placebo on the Brief VisuoSpatial Memory Test Revised (BVMT-R) Total Recall Score.
Description: BVMT-R total recall score. Each of the six equivalent, alternate BVMT-R stimulus forms consists of six geometric figures, printed in a 2 x 3 array, on a separate page of the Recall Stimulus Booklet. In the three Learning Trials, the respondent views the Recall Stimulus page for 10 seconds, then is asked to draw as many of the figures as possible, in their correct page locations. The total recall score is the sum of the three learning trials.
  After a 25-minute delay, which includes primarily verbal activities, the task is repeated. The respondent is asked to identify which of the 12 figures in the Recognition Stimulus Booklet were included in the 6 geometric figures on the original Recall Stimulus page.
  These scores are for the total recall raw score which ranges from 0-36 with 36 being the highest and best possible score.
Time Frame: Baseline, 6 weeks, 12 weeks after beginning Namenda or placebo
Population: All subjects who completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 11 | 11
units on a scale
  baseline score | 18.09 (6.9) | 15.09 (7.8)
  6 week score | 18.18 (7.4) | 17.54 (7.5)
  12 week score | 17.45 (6.8) | 17.18 (8)
Statistical Analysis 1: Comparison: Memantine vs Placebo; Null hypothesis: The change from baseline occurring with memantine is equal to the change from baseline occurring with placebo at 6 weeks for BVMT-R total recall scores; Test type: Superiority or Other; p = 0.34, Sign test — 6 week comparison, alpha = 0.05
Statistical Analysis 2: Comparison: Memantine vs Placebo; Null hypothesis: The change from baseline occurring with memantine is equal to the change from baseline occurring with placebo at 12 weeks for BVLT-R total recall scores; Test type: Superiority or Other; p = 1.0, Sign test — 12 week comparison, alpha = 0.05
Statistical Analysis 3: Comparison: Memantine vs Placebo; Null hypothesis: The change from baseline occurring with memantine is equal to the change from baseline occurring with placebo at 6 weeks for HVLT-R total recall scores; Test type: Superiority or Other; p = 0.54, Wilcoxon (Mann-Whitney) — 6 week comparison, alpha = 0.05
Statistical Analysis 4: Comparison: Memantine vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.91, Wilcoxon (Mann-Whitney) — 12 week comparison, alpha = 0.05

6. Primary Outcome: Improvements From Baseline Scores After 6 and 12 Weeks of Memantine Compared to Placebo on the Brief VisuoSpatial Memory Test Revised (BVMT-R) Delayed Recall Score.
Description: BVMT-R Delayed recall. Each of the six equivalent, alternate BVMT-R stimulus forms consists of six geometric figures, printed in a 2 x 3 array, on a separate page of the Recall Stimulus Booklet. In the three Learning Trials, the respondent views the Recall Stimulus page for 10 seconds, then is asked to draw as many of the figures as possible, in their correct page locations.
  After a 25-minute delay, which includes primarily verbal activities, the task is repeated. The respondent is asked to identify which of the 12 figures in the Recognition Stimulus Booklet were included in the 6 geometric figures on the original Recall Stimulus page.
  These scores are for the delayed recall raw score which ranges from 0 to 12 with 12 being the highest and best possible score.
Time Frame: Baseline, 6 weeks, and 12 weeks after beginning memantine or placebo
Population: All subjects completing the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 11 | 11
units on a scale
  baseline score | 6.64 (3.6) | 6.18 (3.4)
  6 week score | 7.09 (3.8) | 6.27 (3.4)
  12 week score | 7.18 (3.0) | 7.63 (4.0)
Statistical Analysis 1: Comparison: Memantine vs Placebo; Null hypothesis: The change from baseline occurring with memantine is equal to the change from baseline occurring with placebo at 6 weeks for BVMT-R delayed recall scores; Test type: Superiority or Other; p = 0.34, Sign test — 6 week comparison, alpha = 0.05
Statistical Analysis 2: Comparison: Memantine vs Placebo; Null hypothesis: The change from baseline occurring with memantine is equal to the change from baseline occurring with placebo at 12 weeks for BVMT-R delayed recall scores; Test type: Superiority or Other; p = 0.55, Sign test — 12 week comparison, alpha = 0.05
Statistical Analysis 3: Comparison: Memantine vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.37, Wilcoxon (Mann-Whitney) — 6 week comparison, alpha = 0.05
Statistical Analysis 4: Comparison: Memantine vs Placebo; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; p = 0.95, Wilcoxon (Mann-Whitney) — 12 week comparison, alpha = 0.05

7. Secondary Outcome: Improvements From Baseline Scores After 6 and 12 Weeks of Memantine Compared to Placebo on the Symbol Digit Modality Test (SDMT)Written Score.
Description: SDMT Written Scores. SDMT requires the subject to substitute a number for its corresponding geometric figure. There are nine figures. On the record form, there are a series of rows containing geometric figures in the top half, but the bottom half is left blank. When it is clear that the subject understands the task, he or she is told to fill in the remaining boxes as quickly as possible, completing one box at a time, one row at a time, before proceeding to the next. Skipping from box to box with the same geometric figure is not permitted. Subjects receive one point for each correctly completed box. The total score is the total number of correctly completed boxes in the time allowed. The practice items are not counted in the scoring. The test can be administered by having the subject write out the correct response or by having the subject report the correct answer (i.e., number) aloud. Higher scores are better scores and the range of scores can be from 0 to 110 for SDMT written scores.
Time Frame: baseline, 6 weeks, 12 weeks
Population: All subjects completing the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 11 | 11
units on a scale
  baseline score | 35.9 (11.5) | 36.1 (7.9)
  6 week score | 36.5 (9.4) | 39.8 (8.4)
  12 week score | 38.2 (9.8) | 39.8 (7.6)
Statistical Analysis 1: Comparison: Memantine vs Placebo; Null hypothesis: The change from baseline occurring with memantine is equal to the change from baseline occurring with placebo at 6 weeks for the SDMT Written Score; Test type: Superiority or Other; p = 0.75, Sign test — 6 week comparison, alpha = 0.05
Statistical Analysis 2: Comparison: Memantine vs Placebo; Null hypothesis: The change from baseline occurring with memantine is equal to the change from baseline occurring with placebo at 12 weeks for the SDMT Written Score; Test type: Superiority or Other; p = 0.51, Sign test — 12 week comparison, alpha = 0.05
Statistical Analysis 3: Comparison: Memantine vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.31, Wilcoxon (Mann-Whitney) — 6 week comparison, alpha = 0.05
Statistical Analysis 4: Comparison: Memantine vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.46, Wilcoxon (Mann-Whitney) — 12 week comparison, alpha = 0.05

8. Secondary Outcome: Improvements From Baseline Scores After 6 and 12 Weeks of Memantine Compared to Placebo on the Symbol Digit Modality Test (SDMT) Oral Score.
Description: SDMT Oral Score: SDMT requires the subject to substitute a number for its corresponding geometric figure. There are nine figures. On the record form, there are a series of rows containing geometric figures in the top half, but the bottom half is left blank. When it is clear that the subject understands the task, he or she is told to fill in the remaining boxes as quickly as possible, completing one box at a time, one row at a time, before proceeding to the next. Skipping from box to box with the same geometric figure is not permitted. Subjects receive one point for each correctly completed box. The total score is the total number of correctly completed boxes in the time allowed. The practice items are not counted in the scoring. The test can be administered by having the subject write out the correct response or by having the subject report the correct answer (i.e., number) aloud. Higher scores are better scores and the range of scores can be from 0 to 110 for SDMT oral scores.
Time Frame: Baseline, 6 weeks, and 12 weeks after beginning memantine or placebo
Population: All subjects completing the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 11 | 11
units on a scale
  baseline score | 41.1 (12.1) | 41.3 (9.4)
  6 week score | 42.0 (10.3) | 44.1 (6.3)
  12 week score | 43.9 (9.4) | 46.4 (7.3)
Statistical Analysis 1: Comparison: Memantine vs Placebo; Null hypothesis: The change from baseline occurring with memantine is equal to the change from baseline occurring with placebo at 6 weeks for the SDMT Oral Score; Test type: Superiority or Other; p = 0.34, Sign test — 6 week comparison, alpha = 0.05
Statistical Analysis 2: Comparison: Memantine vs Placebo; Null hypothesis: The change from baseline occurring with memantine is equal to the change from baseline occurring with placebo at 12 weeks for the SDMT Oral Score; Test type: Superiority or Other; p = 0.75, Sign test — 12 week comparison, alpha = 0.05
Statistical Analysis 3: Comparison: Memantine vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.37, Wilcoxon (Mann-Whitney) — 6 week comparison, alpha = 0.05
Statistical Analysis 4: Comparison: Memantine vs Placebo; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.45, Wilcoxon (Mann-Whitney) — 12 week comparison, alpha = 0.05

ADVERSE EVENTS:
Time Frame: For each subject, adverse event data was collected during 12 weeks of treatment with memantine, 12 weeks of treatment with placebo, and during 2 separate 3 to 4 week washout periods following the memantine and placebo treatment periods.
Groups:
- Placebo: All 11 subjects completed 12 weeks of placebo treatment. Subjects were given 5 mg per day for 7 days, then 5 mg twice per day for 7 days, then 10 mg AM, 5 mg PM for 7 days, then 10 mg twice daily, as tablet form.
- Memantine: All 11 subjects completed 12 weeks of memantine treatment. Subjects were given 5 mg per day for 7 days, then 5 mg twice per day for 7 days, then 10 mg AM, 5 mg PM for 7 days, then 10 mg twice daily, as tablet form.
- No Treatment (Washout): All 11 subjects completed a 4 week washout between memantine and placebo arms and a 4 week washout at the end of the study.
Arm/Group | Placebo | Memantine | No Treatment (Washout)
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 5/11 | 8/11 | 5/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=11) | Memantine (N=11) | No Treatment (Washout) (N=11)
allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Bilateral calf pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Stomach cramps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3) | 2 (3)
Left great toe nail removed (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Right inguinal strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 2 (2) | 2 (2) | 1 (1)
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Right shoulder strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Left knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Right sided musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Right shoulder muscle strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Left calf strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nervousness (Nervous system disorders) | 0/1 (0) | 1 (1) | 0 (0)
Dry mouth (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Anxiety (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The enrollment goal for the study was 20 subjects. The study included 11 subjects but was terminated due to a lack of additional subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications and Copyrights: INSTITUTE will be free to publish papers dealing with final results of research under this Agreement, 90 days after submitting such papers to FOREST for review providing that INSTITUTE gives due regard to FOREST's comments on the proposed publication.